CLINICAL TRIAL: NCT02147847
Title: Neurological Treatment to Improve the Hearing in Noise Abilities of Older Adults With Hearing Impairments.
Brief Title: Computer-Based Auditory Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Daniel Polley, Assistant Professor in Department of Otology and Laryngology, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-006H-AUD
Record Dates: First submitted 2014-05-15; First posted 2014-05-28 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-05

CONDITIONS: Presbycusis
Keywords: Presbycusis; Hearing In Noise; Hearing Impairment; Hearing Loss; Aging; Plasticity; Video Games; Perceptual Learning
MeSH Terms: conditions — Presbycusis; Hearing Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video game based training 1 (Experimental): Video Game play with training strategy 1
  Interventions: Behavioral: Video game based training 1
- Video game based training 2 (Experimental): Video Game play with training strategy 2
  Interventions: Behavioral: Video game based training 2

INTERVENTIONS:
Behavioral: Video game based training 1 — 32 one-hour, home-based training sessions over 8 weeks
  Arms: Video game based training 1
Behavioral: Video game based training 2 — 32 one-hour, home-based training sessions over 8 weeks
  Arms: Video game based training 2

SUMMARY:
Hearing in noisy environments is a perceptual problem that is ubiquitous in modern industrialized societies. This particular listening context offers a particular challenge to individuals living with hearing impairment (30 million in US alone) even after treatment with hearing aids or cochlear implants. The ability of the brain to extract regularities from the environment and suppress distracting information can be improved with intensive cognitive training. The investigators will test whether the hearing in noise abilities of adults living with hearing impairment can be improved with a cognitive training paradigm.

DETAILED DESCRIPTION:
Hearing impairment (HI) represents the most common cause of moderate to severe disability in the world, with an estimated prevalence of 636 million individuals (30 million in the US alone). Amplification devices (i.e., hearing aids) are commonly used to compensate for HI stemming from acoustic trauma, ototoxic insult, normal aging or other sources of cochlear degeneration. The chief complaint of individuals with HI is hearing in the types of noisy environments that characterize most work, educational, and social situations. Unfortunately, hearing aids do not completely address the perceptual impairments in these situations. That is because the difficulties that individuals with HI have hearing in noise result from the reduced salience of cues that are used to sort out auditory scenes. Making sounds louder improves audibility, but does not afford adaptation of the brain to the abnormal coding of sensory information by the damaged cochlea. The investigators will test whether the hearing in noise abilities of adults living with hearing impairment can be improved with a cognitive training paradigm.

ELIGIBILITY:
Inclusion Criteria:

* Binaural sensorineural hearing impairment
* Use of binaural hearing aids
* Native English Speaker

Exclusion Criteria:

* Significant cognitive impairment
* Significant motor impairment
* History of neurological disease/head trauma
* Use of psychotropic and thyroid medications

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Speech Perception in Noise | up to 3 months
  Participants will report words spoken by a target speaker while several speakers serve as distractors.

SECONDARY OUTCOMES:
Frequency Modulation Detection | up to 3 months
  We will measure the detectability of frequency excursions psychoacoustically.
Stroop Task | up to 3 months
  Participants will be asked to attend and report one feature of a stimulus while ignoring another
Letter-Numbers Sequencing Test | up to 3 months
  Participants are asked to repeat a string of letters and numbers.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Polley, Ph.D., Principal Investigator — Massachusetts Eye and Ear Infirmary, Harvard Medical School
Locations (3):
- United States (3):
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Saint Elizabeth's Medical Center, Brighton, Massachusetts
  - Hudson Valley Audiology Center, New City, New York

REFERENCES:
- [Background] Anderson S, White-Schwoch T, Parbery-Clark A, Kraus N. Reversal of age-related neural timing delays with training. Proc Natl Acad Sci U S A. 2013 Mar 12;110(11):4357-62. doi: 10.1073/pnas.1213555110. Epub 2013 Feb 11. PMID 23401541
- [Background] Keeling MD, Calhoun BM, Kruger K, Polley DB, Schreiner CE. Spectral integration plasticity in cat auditory cortex induced by perceptual training. Exp Brain Res. 2008 Feb;184(4):493-509. doi: 10.1007/s00221-007-1115-9. Epub 2007 Sep 21. PMID 17896103
- [Background] Polley DB, Heiser MA, Blake DT, Schreiner CE, Merzenich MM. Associative learning shapes the neural code for stimulus magnitude in primary auditory cortex. Proc Natl Acad Sci U S A. 2004 Nov 16;101(46):16351-6. doi: 10.1073/pnas.0407586101. Epub 2004 Nov 8. PMID 15534214
- [Background] Polley DB, Steinberg EE, Merzenich MM. Perceptual learning directs auditory cortical map reorganization through top-down influences. J Neurosci. 2006 May 3;26(18):4970-82. doi: 10.1523/JNEUROSCI.3771-05.2006. PMID 16672673
- [Background] Li RW, Ngo C, Nguyen J, Levi DM. Video-game play induces plasticity in the visual system of adults with amblyopia. PLoS Biol. 2011 Aug;9(8):e1001135. doi: 10.1371/journal.pbio.1001135. Epub 2011 Aug 30. PMID 21912514
- [Background] Sweetow RW, Sabes JH. The need for and development of an adaptive Listening and Communication Enhancement (LACE) Program. J Am Acad Audiol. 2006 Sep;17(8):538-58. doi: 10.3766/jaaa.17.8.2. PMID 16999250
- [Background] Bao S, Chang EF, Woods J, Merzenich MM. Temporal plasticity in the primary auditory cortex induced by operant perceptual learning. Nat Neurosci. 2004 Sep;7(9):974-81. doi: 10.1038/nn1293. Epub 2004 Aug 1. PMID 15286790
- [Background] Green CS, Bavelier D. Action video game modifies visual selective attention. Nature. 2003 May 29;423(6939):534-7. doi: 10.1038/nature01647. PMID 12774121
- [Background] Green CS, Pouget A, Bavelier D. Improved probabilistic inference as a general learning mechanism with action video games. Curr Biol. 2010 Sep 14;20(17):1573-9. doi: 10.1016/j.cub.2010.07.040. PMID 20833324
- [Background] Deveau J, Ozer DJ, Seitz AR. Improved vision and on-field performance in baseball through perceptual learning. Curr Biol. 2014 Feb 17;24(4):R146-7. doi: 10.1016/j.cub.2014.01.004. No abstract available. PMID 24556432
- [Background] Li J, Thompson B, Deng D, Chan LY, Yu M, Hess RF. Dichoptic training enables the adult amblyopic brain to learn. Curr Biol. 2013 Apr 22;23(8):R308-9. doi: 10.1016/j.cub.2013.01.059. PMID 23618662
- [Background] Lim SJ, Holt LL. Learning foreign sounds in an alien world: videogame training improves non-native speech categorization. Cogn Sci. 2011 Sep-Oct;35(7):1390-405. doi: 10.1111/j.1551-6709.2011.01192.x. Epub 2011 Aug 9. PMID 21827533
- [Background] Merzenich MM, Jenkins WM, Johnston P, Schreiner C, Miller SL, Tallal P. Temporal processing deficits of language-learning impaired children ameliorated by training. Science. 1996 Jan 5;271(5245):77-81. doi: 10.1126/science.271.5245.77. PMID 8539603
- See also: Laboratory website of Principal Investigator — http://scholar.harvard.edu/polleylab